CLINICAL TRIAL: NCT01811849
Title: A Double-blind Study of the Pharmacokinetic Properties of BIOD-238 and BIOD-250 Compared to Humalog® in Subjects With Type 1 Diabetes Including Assessments of Safety and Injection Site Toleration
Brief Title: Pharmacokinetic and Injection Site Toleration of BIOD-238 and BIOD-250 Compared to Humalog® in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4-102
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- BIOD-238 (Experimental): Subcutaneous injection
  Interventions: Drug: Insulin LISPRO
- BIOD-250 (Experimental): Subcutaneous injection
  Interventions: Drug: Insulin LISPRO
- Humalog (Active Comparator): Subcutaneous injection
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: Insulin LISPRO
  Arms: BIOD-238
Drug: Insulin LISPRO
  Arms: BIOD-250
Drug: Insulin LISPRO
  Arms: Humalog

SUMMARY:
A Double-blind Study of the Pharmacokinetic Properties of BIOD-238 and BIOD-250 Compared to Humalog® in Subjects with Type 1 Diabetes

DETAILED DESCRIPTION:
The purpose of this study is to assess the speed of absorption of BIOD-238 and BIOD-250 compared to Humalog®. Secondary objectives are to assess other pharmacokinetic characteristics of BIOD-238 and BIOD-250 compared to Humalog®, and to evaluate the safety and tolerability of BIOD-238 and BIOD-250 compared to Humalog®.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 to ≤70 years
* Body Mass Index: ≥18 and ≤35 kg/m2
* Diagnosed with Type 1 Diabetes Mellitus for at least 1 year

Exclusion Criteria:

* Type 2 diabetes mellitus
* Serum C-peptide >1.0 ng/mL
* HbA1c >10.0%
* History of hypersensitivity to any of the components in the study medication
* Treatment with any other investigational drug in the last 30 days before dosing.
* Current drug or alcohol abuse, or a history of drug or alcohol abuse which in the opinion of the Investigator will impair subject safety, protocol compliance, or interpretation of study results. Caffeine, nicotine or alcohol addiction which might be expected to result in withdrawal symptoms during the course of a study dosing day would fall into this category.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to 1/2 maximal insulin concentration | 480 minutes

SECONDARY OUTCOMES:
Time to maximal insulin concentration | 480 minutes
Time to 1/2 maximal insulin concentration after peak | 480 minutes
Visual analog scale | 30 minutes
AUC 0-30 and AUC 0-60 | 60 minutes